CLINICAL TRIAL: NCT02598830
Title: The Granheim COPD Study: Effects of Vitamin D3-supplementation on the Efficacy of Strength Training in COPD Patients and Healthy Controls - a Double-blinded RCT
Brief Title: The Granheim COPD Study - Vitamin D and Strength Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inland Norway University of Applied Sciences (Other)
Collaborators: Sykehuset Innlandet HF (Other); Lillehammer Hospital for Rheumatic Diseases (Other); University of Bergen (Other); University of Copenhagen (Other); Norwegian School of Sport Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Trainsome 2014#004
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Cachexia; Vitamin D; Muscle; Strength training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cachexia | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3+str.training, COPD & Healthy (Experimental): Vitamin D3 capsules for 30 weeks:
  * weeks 1-2: 10000 IU/day (equivalent to 250 ug), accompanied by 1000 mg Ca2+
  * weeks 3-30: 2000 IU/day (equivalent to 50 ug), accompanied by 1000 mg Ca2+
  Progressive unilateral strength training of the legs for 3+10 weeks (weeks 15-28); leg 1 = high-load training, leg 2 = low-load training, allocated to left and right foot in a randomized manner:
  * weeks 15-17, familiarization period
  * week 18, test period
  * weeks 19-28, intervention period
  * weeks 29-30, test period
  Interventions: Dietary Supplement: Vitamin D3
- Placebo+str.training, COPD & Healthy (Placebo Comparator): Placebo capsules for 30 weeks (the number of capsules ingested each day match those of the vitamin D3 group)
  Progressive unilateral strength training of the legs for 3+10 weeks (weeks 15-28); leg 1 = high-load training, leg 2 = low-load training, allocated to left and right foot in a randomized manner:
  * weeks 15-17, familiarization period
  * week 18, test period
  * weeks 19-28, intervention period
  * weeks 29-30, test period
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 dissolved in olive oil, encapsuled
  Other Names: cholecalciferol
  Arms: Vitamin D3+str.training, COPD & Healthy
Dietary Supplement: Placebo — Olive oil, encapsuled
  Arms: Placebo+str.training, COPD & Healthy

SUMMARY:
This study evaluates the effect of vitamin D supplementation on outcomes of 10 weeks progressive strength training in 100 ageing subjects (>45 years of age). Participants will be recruited into two similarly sized strata; one containing COPD patients and one containing healthy subjects of similar age. In each stratum, half the participants will receive vitamin D supplementation and half the participants will receive placebo

DETAILED DESCRIPTION:
Physical activity is a potent way of relieving some of the adverse morbidities associated with COPD, such as muscle atrophy and reduced muscle quality. It is thus problematic that 20-30% of patients fail to elicit positive adaptations to training. This oddity has been ascribed inherent muscular properties, with potential links to comorbidities such as vitamin D and testosterone deficiency and the nature of the training program. In the present project, a double-blinded RCT will be performed to disclose the functional and biological efficacy of vitamin D supplementation (with concomitant ingestion of 1000 mg Ca2+) on the outcomes of 10 wks strength training in 100 aging individuals with or without COPD. The strength training intervention will be preceded by 3 weeks of progressive introduction to training protocols.

50 COPD patients and 50 healthy subjects will be allocated into two strata and separately randomized into two equally sized supplementation groups; (1) vitamin D3 and (2) placebo. The planned 50:50 ratio between COPD patients and healthy individuals may change, depending on the access to COPD patients. All subjects will perform lower-limb strength-training protocols in a contralateral manner: (leg 1) high-resistance (10 RM) and (leg 2) low-resistance (30 RM). Such a one-limb-at-a-time protocol ensures training that is unconfined by the cardiorespiratory limitations inherent to these patients, and allow comparison of the two training modalities in a manner unconfined by individual variation in exercise adaptability. A pilot study investigating the possible central pulmonary capacity limitation to two-legged strength training exercise in COPD patients will be performed. In this pilot study, we will compare exercise performance involving large and small muscle mass. In addition, all subjects will perform a selection of bilateral upper body exercises (10 RM), ensuring adequate hormonal responses and compliance to the study. The study is likely to revitalize guidelines for rehabilitation of COPD patients, and to provide vital information regarding the role of vitamin D in adaptations to strength training.

For outcome measures specific to COPD pasients, final analyses will be performed on data from the COPD population only. For other outcome measures, final analyses will be performed on data merged from COPD patients and healthy subjects. An important rationale behind implementing healthy control subjects is to increase the statistical power of outcome measures unrelated to COPD epidemiology, which are of general relevance to physiological adaptation to strength training. In a related set of analyses, we will perform between-groups comparisons, including multivariate analyses. We will also compare the efficacy of high- and low-resistance strength training in COPD patients and healthy control subjects. The two training modalities are expected to result in similar muscular adaptations.

In general, baseline vitamin D levels in blood, measured as 25(OH)D, is anticipated to be a determinant of the efficacy of the strength training intervention. In response to vitamin D3 supplementation, individuals with low baseline levels of 25(OH)D are expected to display more pronounced changes in biological active vitamin D, leading to more pronounced changes in functional and biological outcome measures in response to strength training. In contrast, supplementation may not lead to further elevation of blood 25(OH)D levels in individuals with high baseline levels, essentially meaning that vitamin D3 ingestion will be leveled out by or exceeded by the elimination of vitamin D derivatives. In these individuals, vitamin D3 ingestion will not have an additive effect on functional and biological outcome measures in response to strength training. To assess individual variation in vitamin D responses, data on functional and biological variables will be divided into quartiles based on baseline 25(OH)D-levels, whereupon comparisons will be made between low-end and high-end quartiles. Individual variation in responses to vitamin D supplementation and strength training will also be assessed using a mixed model approach.

ELIGIBILITY:
COPD group

Inclusion Criteria:

* Stable COPD at GOLD stage II or III, FEV1/FVC < 0.7 and FEV1 <80% and >30% of predicted
* >45 years of age

Exclusion Criteria:

* Unstable cardiovascular disease
* Chronic granulomatous
* Known active malignant disease within last 5 years
* Physically disabling muscloskeletal diseases
* Peroral use of steroids within last 2 months
* Serious psychiatric comorbidity
* Less than 4 weeks since last return t o habit ual condit ion from exacerbation
* Failing to understand Norwegian literary or verbally
* Medical record diagnosis of asthma
* More than one bout of strength training per week during the last 6 months leading up to the project

Healthy control group

Inclusion Criteria:

- >45 years of age

Exclusion Criteria:

* COPD
* Unstable cardiovascular disease
* Chronic granulomatous
* Known active malignant disease within last 5 years
* Physically disabling muscloskeletal diseases
* Peroral use of steroids within last 2 months
* Serious psychiatric comorbidity
* Failing to understand Norwegian literary or verbally
* Medical record diagnosis of asthma
* More than one bout of strength training per week during the last 6 months leading up to the project

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Muscle size | Changes from before to after the strength training intervention (week 19 to week 28)
  Muscle cell cross-sectional area measured in biopsies from m. vastus lateralis using immunohistochemistry
Muscle phenotype | Changes from before to after the strength training intervention (week 19 to week 28)
  Muscle fiber type composition measured in biopsies from m. vastus lateralis using immunohistochemistry

SECONDARY OUTCOMES:
Lung function | Changes from before to after the strength training intervention (week 19 to week 28)
  Lung function measured using spirometry
One-legged cycling | Changes from before to after the strength training intervention (week 19 to week 28)
  Performance indicies measured during an incremental one-legged cycling test
Hormones in blood | Changes over the course of the intervention (week 0 to 28)
  Levels of hormones in blood
Cytokines in blood | Changes over the course of the intervention (week 0 to 28)
  Levels of cytokines in blood
Steroids in skeletal muscle | Changes over the course of the intervention (week 0 to 28)
  Levels of steroids in m. vastus lateralis
Androgen-converting enzymes in skeletal muscle | Changes from before to after the strength training intervention (week 19 to week 28)
  Levels of androgen-converting enzymes in m. vastus lateralis
Gene expression in skeletal muscle | Changes from before to after the strength training intervention (week 19 to week 28)
  RNA (e.g. messenger RNA, ribosomal RNA, microRNA, long non-coding RNA) abundances in m. vastus lateralis, measured both as single genes and at the level of the transcriptome
Gene expression in skeletal muscle | Changes from before to after familiarization to strength training (week 15 to week 17)
  RNA (e.g. messenger RNA, ribosomal RNA, microRNA, long non-coding RNA) abundances in m. vastus lateralis, measured both as single genes and at the level of the transcriptome
Protein abundances in skeletal muscle | Changes from before to after the strength training intervention (week 19 to week 28)
  Levels of proteins and their modification status (e.g. phosphorylation) in m. vastus lateralis, measured at the level of single proteins and at the level of the proteome
Protein abundances in skeletal muscle | Changes from before to after familiarization to strength training (week 15 to week 17)
  Levels of proteins and their modification status (e.g. phosphorylation) in m. vastus lateralis, measured at the level of single proteins and at the level of the proteome
Vitamin D in blood | Changes over the course of the intervention (week 0 to 28)
  Levels of vitamin D in blood
Step test | Changes from before to after the strength training intervention (week 19 to week 28)
  Performance and performance indicies measured during a 6 minutes step test
Pasient-reported outcome measures, generic | Changes from before to after the strength training intervention (week 19 to week 28)
  Pasient-related outcome measures assessed using the generic survey SF-36
Pasient-reported outcome measures, COPD-specific | Changes from before to after the strength training intervention (week 19 to week 28)
  COPD-specific pasient-reported outcome assessed using COPD assessment test
Body mass composition | Changes from before to after the strength training intervention (week 19 to week 28)
  Body mass composition measured using Dual-energy X-ray absorptiometry (DXA)
Bilateral upper body maximal strength | Changes from before to after the strength training intervention (week 19 to week 28)
  The ability of muscles of the upper body to exert maximal force during dynamic movements
Grip strength | Changes from before to after the strength training intervention (week 19 to week 28)
  Isometric hand grip strength
Sit-to-stand test | Changes from before to after the strength training intervention (week 19 to week 28)
  Performance and performance indicies measured during a sit-to-stand test
Unilateral lower body maximal muscle strength | Changes from before to after the strength training intervention (week 19 to week 28)
  The ability of muscles of the lower body to exert maximal force during dynamic movements
Unilateral lower body muscle endurance | Changes from before to after the strength training intervention (week 19 to week 28)
  The ability of muscles of the lower body to perform repeated dynamic contractions at a specified submaximal load to exhaustion
Bilateral upper body muscle endurance | Changes from before to after the strength training intervention (week 19 to week 28)
  The ability of muscles of the upper body to perform repeated dynamic contractions at a specified submaximal load to exhaustion
Unilateral lower body isokinetic muscle strength | Changes from before to after the strength training intervention (week 19 to week 28)
  The ability of muscles of the lower body to exert maximal force during isokinetic movements
Daily life activity level | Changes from before to after the intervention (week 0 to week 28)
  Daily life activity level measured using accelerometer
Muscle cell biological traits | Changes from before to after the strength training intervention (week 19 to week 28)
  Muscle cell biological traits, including numbers of myonuclei, satelitte cells and capillaries, measured in biopsies from m. vastus lateralis using immunohistochemistry
Muscle mitochondrial quantities | Changes from before to after the strength training intervention (week 19 to week 28)
  Mitochondrial quantities measured in biopsies from m. vastus lateralis
Muscle mitochondrial functions | Changes from before to after the strength training intervention (week 19 to week 28)
  Mitochondrial functions measured in biopsies from m. vastus lateralis

OTHER OUTCOMES:
Training diary | Measured over the course of the strength training familiarization period and the strength training intervention (week 15 to week 28)
  Training diary containing information about type of training, duration of training and training intensity
Dietary registration | Registred at one time point during the strength training intervention (~week 23, registred over four days)
  Detailed registration of food intake
Self-reported information on lifestyle-related aspects | Measured over the course of the intervention (week 0 to week 28)
  Disease, symptoms, injury, vitamin D-intake, time spent outdoors, solarium, training background, smoking, etc

CONTACTS AND LOCATIONS:
Overall Officials: Knut Sindre Mølmen, MSc, Principal Investigator — Inland Norway University of Applied Sciences
Locations (1):
- Inland Norway University of Applied Sciences, Lillehammer, Norway

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to the academic community through the general biobank "The Trainsome - effects of exercise and environment on human cells" (REK-2013/2045, Regional Comitees for Medical and Health Research Ethics South East). Data will be available on request and will be restricted to scientists and/or projects with a sound scientific purpose and rationale.

REFERENCES:
- [Derived] Molmen KS, Hammarstrom D, Falch GS, Grundtvig M, Koll L, Hanestadhaugen M, Khan Y, Ahmad R, Malerbakken B, Rodolen TJ, Lien R, Ronnestad BR, Raastad T, Ellefsen S. Chronic obstructive pulmonary disease does not impair responses to resistance training. J Transl Med. 2021 Jul 6;19(1):292. doi: 10.1186/s12967-021-02969-1. PMID 34229714